CLINICAL TRIAL: NCT05257616
Title: Effect of Cervical Mobility on Cardiovascular And Respiratory Outcomes Among Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Zoya 048-538
Record Dates: First submitted 2021-11-05; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain; Blood Pressure
Keywords: Neck pain; Blood pressure; Heart rate; Range of motion; Respiratory rate
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: It include the control and experimental group.
Who Masked: Participant
Masking Description: The participant were blinded to the both treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Questionnaires were given to the participants. Before the initiation of treatment, procedure and consent details were explained and verbally translated into the native languages of participants, followed by the written signed approval on the questionnaire. Cervical ranges were measured using inclinometer which included neck flexion, extension, left and right side bending. Succeeding it were vitals in which oxygen saturation, heart rate, blood pressure, ventilation rate were jotted along with pain measurement using NPRS scale.
  Interventions: Other: Traction Mobilization technique
- Experimental Group (Active Comparator): Questionnaires were given to the participants. Before the initiation of treatment, procedure and consent details were explained and verbally translated into the native languages of participants, followed by the written signed approval on the questionnaire. Cervical ranges were measured using inclinometer which included neck flexion, extension, left and right side bending. Succeeding it were vitals in which oxygen saturation, heart rate, blood pressure, ventilation rate were jotted along with pain measurement using NPRS scale.
  Interventions: Other: Traction Mobilization technique with SNAGS

INTERVENTIONS:
Other: Traction Mobilization technique — Traction Mobilization was given by Researcher at the cervical spine followed by a one minute interval before post vitals were taken, that marked the end of the first session. Three similar sessions succeeded the first, each at an interval of 2 days for 2 weeks between the first and second session; third and fourth session respectively. At the end of the fourth session, cervical ranges and pain intensity were noted again. Participant sits comfortably or leans against a chair backrest. Palms of the hands are placed on the mastoid processes of the patient's skull while pressing the elbows in a caudal direction. It was held for 5 seconds then relaxed.
  Arms: Control Group
Other: Traction Mobilization technique with SNAGS — Traction Mobilization with SNAGS were given at the cervical spine followed by a one minute interval before post vitals were taken, that marked the end of the first session. Three similar sessions succeeded the first, each at an interval of 2 days for 2 weeks between the first and second session; third and fourth session respectively. At the end of the fourth session, cervical ranges and pain intensity were noted again The position of the therapist is behind him or her, medial border of therapist's right thumb is used to contact the spinous process of C6 vertebrae i.e. level above the suspected painful or hypo mobile region. Therapist's left thumb reinforces his/her (right) contact thumb. Therapist fingers are gently placed along the patient's mandible or thorax. Following the treatment plane towards the eye, lift comes from the mobilizing thumb not the contact thumb. While the glide is maintained, the patient is asked to rotate his/her head towards the side of pain or hypo mobility.
  Arms: Experimental Group

SUMMARY:
In some individuals, neck pain subsides within a year but reappearance is surpassing while for some patients it prevails for lifetime. According to a study on global burden of disease performed in 2010, neck pain was rated as number 4th when measured with Years Lived With Disability (YLDs) and stood 21st when overall burden was concerned. The estimated 1 year incidence of neck pain from available studies ranges between 10.4% and 21.3% with a higher incidence noted in office and computer workers. While the overall prevalence of neck pain in the general population ranges between 0.4% and 86.8% ; point prevalence ranges from 0.4% to 41.5% and 1 year prevalence ranges from 4.8% to 79.5%. Occurrence of neck pain is generally higher in women, high-income countries compared with low- and middle-income countries and in urban areas compared with rural areas. In addition, the patient characteristics like psychosocial factors are determinants, risk factors and prognostic factors of neck pain but this knowledge doesn't provide adequate information to the physician to deal with such patients.

DETAILED DESCRIPTION:
Neck pain is the sense of discomfort that could be felt in the cervical and upper thoracic region. It's an ubiquitous human perception. Non-specific neck pain has a postural or mechanical basis and affects about two thirds of people at some stage, especially in the middle age. Acute neck pain resolves within days or weeks, but may become chronic in about 10% of people. Many individuals have asymptomatic neck pain due to various hidden pathologies and improper postural characteristics which is only noticeable after detailed screening and scans.

Heart and lungs are the main organs housed by the thoracic cage with all their vascular and nervous supply passing through the cervical and the thoracic spine. The respiratory system could be affected by the musculoskeletal system of the body. As there are accessory respiratory muscles of respiration that are attached to the neck, chest wall and/or abdomen.

Bad posture, for instance, can lead to reduction in power of the neck muscles hence reducing power of the respiratory muscles creating negative effect on the thoracic expansion, alveolar ventilation, reducing lung volume and vital capacity.

Every health system is indicated by certain measures, vital signs are indicative of the health of cardiovascular and respiratory system as well as body as a whole. These physiological observations generally include blood pressure (BP), heart rate (HR), and ventilation rate (VR), temperature (Temp), and oxygen saturation (SPO2) in the blood. Another vital sign, known as the fifth vital sign is Pain.

Changes or deviation of the vital signs from its normal ranges help evaluate and manage any adverse event such as cardiac arrest or sudden death and help in preventing many such deadly events by early recognition and prompt treatments and also help reduce mortality and morbidity.

Several studies have been known to show that alterations in vital signs are not only seen as a result of any pathological event but also any non-pathological as well. Any type of physiological movements of body part such as the spine as a whole or interventional movements, several exercises, mobilization or manipulations, to any segment of the spine like cervical, thoracic or lumbar, have a specific effect on the vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Cervical pain
* Cervical hypo mobility

Exclusion Criteria:

* History of cervical trauma or injury
* Any structural deformity
* Vertebral instability
* Cardiac and respiratory complications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-03-11 (Estimated)

PRIMARY OUTCOMES:
Cardiac outcome | 4 weeks
  Heart rate was measured by using handheld oximeter as beats per min
Respiratory outcome | 4 weeks
  Respiratory Rate was calculated by thoraco-abdominal expansion and it was denoted as respiratory rate per minute
Vascular Outcome | 4 weeks
  Blood pressure was measured by using sphygmanometer in mmHg
Oxygen Saturation | 4 weeks
  Oxygen saturation was noted by using pulse oximeter

SECONDARY OUTCOMES:
Range of motion of cervical spine | 4 weeks
  cervical flexion, extension, left and right side bending via inclinometer
Numeric Pain Rating Scale | 4 weeks
  Pain was assessed before and after treatment using Numeric pain rating scale. this scale has minimum score of 0 and o indicates no pain whereas 10 is the maximum score of scale which shows worst pain ever by using nprs.

CONTACTS AND LOCATIONS:
Overall Officials: Zoya Mehmood, MS-OMPT, Principal Investigator — Shifa tameer e millat university Islamabad
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll LJ, Hogg-Johnson S, van der Velde G, Haldeman S, Holm LW, Carragee EJ, Hurwitz EL, Cote P, Nordin M, Peloso PM, Guzman J, Cassidy JD. Course and prognostic factors for neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S87-96. doi: 10.1016/j.jmpt.2008.11.013. PMID 19251079
- [Background] Braun BL. Postural differences between asymptomatic men and women and craniofacial pain patients. Arch Phys Med Rehabil. 1991 Aug;72(9):653-6. PMID 1859260
- [Background] Schellhas KP, Smith MD, Gundry CR, Pollei SR. Cervical discogenic pain. Prospective correlation of magnetic resonance imaging and discography in asymptomatic subjects and pain sufferers. Spine (Phila Pa 1976). 1996 Feb 1;21(3):300-11; discussion 311-2. doi: 10.1097/00007632-199602010-00009. PMID 8742205
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Blozik E, Laptinskaya D, Herrmann-Lingen C, Schaefer H, Kochen MM, Himmel W, Scherer M. Depression and anxiety as major determinants of neck pain: a cross-sectional study in general practice. BMC Musculoskelet Disord. 2009 Jan 26;10:13. doi: 10.1186/1471-2474-10-13. PMID 19171034
- [Background] Kim SY, Kim NS, Kim LJ. Effects of cervical sustained natural apophyseal glide on forward head posture and respiratory function. J Phys Ther Sci. 2015 Jun;27(6):1851-4. doi: 10.1589/jpts.27.1851. Epub 2015 Jun 30. PMID 26180334
- [Background] Walid MS, Donahue SN, Darmohray DM, Hyer LA Jr, Robinson JS Jr. The fifth vital sign--what does it mean? Pain Pract. 2008 Nov-Dec;8(6):417-22. doi: 10.1111/j.1533-2500.2008.00222.x. Epub 2008 Jul 25. PMID 18662363 (Retraction: PMID 19400820 Pain Pract. 2009 May-Jun;9(3):245)
- [Background] Noten S, Meeus M, Stassijns G, Van Glabbeek F, Verborgt O, Struyf F. Efficacy of Different Types of Mobilization Techniques in Patients With Primary Adhesive Capsulitis of the Shoulder: A Systematic Review. Arch Phys Med Rehabil. 2016 May;97(5):815-25. doi: 10.1016/j.apmr.2015.07.025. Epub 2015 Aug 15. PMID 26284892
- [Background] Hearn A, Rivett DA. Cervical SNAGs: a biomechanical analysis. Man Ther. 2002 May;7(2):71-9. doi: 10.1054/math.2002.0440. PMID 12151243
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284